CLINICAL TRIAL: NCT06666803
Title: Functional, Personalised and Integrated Profiling of Biopsied Pancreatic Tumours
Brief Title: Functional, Personalised and Integrated Profiling of Biopsied Pancreatic Tumours (CancerProfile by FNB)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Collaborators: Luxembourg Institute of Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-003; 2024-A00903-44 (Other: ANSM)
Record Dates: First submitted 2024-10-23; First posted 2024-10-31 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma
Keywords: PDAC; EUS; FNB; PDO; organoid; OCT
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FNB and blood sample analysis (Experimental)
  Interventions: Other: FNB sampling; Biological: blood sampling

INTERVENTIONS:
Other: FNB sampling — A supplementary FNB will be performed during the EUS procedure. Sample will be processed to obtain organoids and assess their morphological, proliferative and genetics characteristics.
Biological: blood sampling — A blood withdrawal will be performed during the EUS procedure. Sample will be processed to assess organoids morphological, proliferative and genetics characteristics.

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC) has the poorest prognosis of all digestive cancers due to lack of early diagnosis and limited response to treatment. Patient-derived organoid technology has become a mainstay of precision oncology, enabling personalised functional characterisation of tumours (e.g. treatment evaluation and drug screening). Initial research carried out as part of the Cancer Profile project has produced the first organoids from resected PDAC parts.

Only 15-20% of patients can benefit from surgical resection, which remains the only curative treatment. In contrast, most patients with PDAC undergo diagnostic fine-needle biopsies (FNB) using an echo-endoscopic procedure (EUS). The next step is therefore the reliable generation of organoids from limited quantities of biopsy material obtained by 'EUS-FNB'.

The aim of the study presented here is to validate these organoids on the basis of the following characteristics: (i) morphological and proliferative characteristics, (ii) recapitulation of the genetic characteristics of the original tumour, (iii) expression of tumour markers.

DETAILED DESCRIPTION:
Pancreatic Ductal AdenoCarcinoma (PDAC) has the poorest prognosis of all digestive cancers due to lack of early diagnosis and limited response to treatment. Its mortality rate is expected to increase in Western countries as populations age and obesity levels rise. Its diagnosis is generally made late in the course of the disease and only 15-20% of patients can benefit from surgical resection, which remains the only curative treatment. Thus, palliative chemotherapy remains a mainstay of the management of this disease. Despite the new approach to treating advanced cancers using molecular characterisation of tumour tissue, only a small subset of patients has access to this personalised treatment and around 13% of patients show a significant response.

Patient-derived organoid (PDO) technology enables personalised functional characterisation of tumours (e.g. treatment evaluation and drug screening).

PDO are created from adult tumour-derived stem cells and self-organise into structures similar to the corresponding tissue architecture in vivo. In pancreatic cancer, PDO have recapitulated the histology and genetic alterations of the original tumour and have been proved reliable in predicting sensitivities to a range of therapeutic compounds. While the majority of PDAC organoids described have been created from surgical resections, only a few examples of PDAC organoids successfully generated from biopsies have been reported.

Given that most PDAC patients are not eligible for surgical resection and therefore undergo diagnostic fine-needle biopsies (FNB) by endoscopic ultrasound (EUS) (EUS-FNB), efforts are needed to improve the generation of PDAC organoids from limited quantities of material. This will ensure that as many PDAC patients as possible can benefit from large-scale drug screening, a technic able to validate gene-drug associations, guide treatment decision-making and known to be well-suited to PDO.

The Cancer Profile project is a European collaboration between the IHU Strasbourg and the LIH, funded respectively by the ANR (Agence Nationale de la Recherche, France) and the FNR (Fonds National de la Recherche, Luxembourg). Its ultimate aim is to be able to profile each tumour sample accurately, in an automated and personalised way. A first trial has enabled the establishment of the technique and conditions for culturing spheroids of pancreatic origin.

The study proposed here is the next step in this project: the reliable generation of organoids from limited quantities of biopsy material obtained by EUS-FNB. This routine procedure is mandatory in the PDAC standard care to obtain tumour tissue for minimally invasive diagnosis and preoperative procedures such as preoperative chemotherapy.

In this clinical study, one to two biopsies will be devoted to the usual analysis performed as part of the care, and a supplementary biopsy will be added for the protocol. This biopsy will be divided in three parts: (i) a sample will be send for organoid culture, (ii) a sample will be preserved in liquid nitrogen and analysed later to check whether the mutations observed in the organoid are indeed identical to those present in the initial tissue, (iii) and a third sample will be analysed by Dynamic Full-field Optical coherence tomography (D-FF-OCT), an innovative technique for imaging living tissue. A blood sample will also be withdrawn for genomic analysis.

Once the first organoids are obtained, they will be validated on the basis of the following characteristics: (i) morphological and proliferative characteristics, (ii) genetic characteristics, and (iii) expression of tumour markers.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient over 18 years of age.
* Patient undergoing echo-endoscopy with certainty/suspicion of fine needle biopsy (EUS-FNB).
* Suspicion of pancreatic lesion
* Patient able to receive and understand information relating to the research protocol and to give consent.
* Patient affiliated to the French social security system.

Exclusion Criteria:

* Patient not programmed for endoscopy with certainty/suspicion of fine needle biopsy (EUS-FNB).
* Patient undergoing echo-endoscopy and presenting a high risk that may prevent EUS-FNB.
* Patient with degenerated Intraductal papillary mucinous neoplasm (IPMN)
* Patient with acute pancreatitis within 4 weeks prior to EUS
* Pregnant or breast-feeding patient
* Patient under court protection.
* Patient under guardianship or curatorship.
* Patient in a situation of social vulnerability.
* Patient under legal protection or unable to express his/her opposition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Organoid culture from PDAC EUS-FNB biopsy | 8 weeks
  Qualitative assessment in the obtention of organoids. The main objective will be validated when a culture of functional organoids is generated.

SECONDARY OUTCOMES:
Evaluation of the protocol for culturing organoids derived from PDAC EUS-FNB biopsies. | 3 months
  Evaluation of the mutations found in the organoid from the EUS-FNB biopsies compared to those in the original sample preserved in liquid nitrogen (qualitative criterion).
Evaluation of the protocol for culturing organoids derived from PDAC EUS-FNB biopsies. | 3 months
  Evaluation of the mutations observed in the cancerous tissue (snap-frozen sample) compared to those observed in the blood sample from the same patient.
Assessment of the overall accuracy of characterising PDAC EUS-FNB samples by optical slicing based on dynamic full-field optical coherence tomography (D-FF-OCT) | Day 1
  Number of EUS-FNB tumour samples confirmed by D-FF-OCT, compared with the total number of samples taken.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of hepato-gastroenterology, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No